CLINICAL TRIAL: NCT06129279
Title: Examining the Effect of Emotional Freedom Technique on Quality of Life and Symptoms in Dysmenorrhea
Brief Title: Effect of Emotional Freedom Technique on Symptoms in Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Ayse Cuvadar, Assistant Professor, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: E-77192459-050.99-232650
Record Dates: First submitted 2023-11-04; First posted 2023-11-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Woman; Pain
Keywords: dysmenorrhea; woman; quality of life
MeSH Terms: conditions — Pain; Dysmenorrhea

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention (EFT) group (Experimental): In order to determine the students who meet our study criteria, PİF, DDF, VAS, MSS and Short Form 36 will be applied for the pre-test to female students studying in the relevant departments of KBÜ SBF.
  To EFT Group; After the first tests are done, the 1st EFT session will be held, the 2nd EFT session will be held 30 days later, and the final tests will be done 30 days later. During this period, affirmations will be given depending on the need. Each session is planned to last an average of 45 minutes - 1 hour, and duration and affirmations will be arranged according to the woman's individual difficulties, perspective, support systems, past traumas and emotional blockages.
  4th Procedure: Preliminary tests will be carried out and then the 1st EFT session will be held.
  5. Procedure: After 30 days, the first final tests will be performed and then the second EFT session will be held.
  Procedure 6: After 30 days, only the 2nd final tests will be performed.
  Interventions: Other: EFT group
- Control group (No Intervention): In order to determine the students who meet our study criteria, PİF, DDF, VAS, MSS and Short Form 36 will be applied for the pre-test to female students studying in the relevant departments of KBÜ SBF. Students in the control group will receive routine counseling regarding primary dysmenorrhea, and no extra intervention or practice will be performed.
  Procedure 1: Preliminary tests will be conducted and then general training for dysmenorrhea will be conducted.
  2nd Process: 30 days later, the questions of the students who will take the 1st post-test will be answered.
  3rd Procedure: After 30 days, the second final tests will be performed.

INTERVENTIONS:
Other: EFT group — Preliminary tests will be carried out and then the 1st EFT session will be held.
  After 30 days, the first final tests will be performed and then the second EFT session will be held.
  After 30 days, only the 2nd final tests will be performed.
  Arms: İntervention (EFT) group

SUMMARY:
1. Reducing symptoms with EFT in young women suffering from dysmenorrhea
2. Improving the quality of life of young women suffering from dysmenorrhea
3. Raising women's awareness for EFT
4. Reducing healthcare costs for dysmenorrhea

DETAILED DESCRIPTION:
Primary dysmenorrhea, the most common form of dysmenorrhea, is a problem characterized by pain that begins in the lower abdomen before or with menstruation, lower back pain and pain radiating to the legs. The Emotion Freedom Techniqu has become a manualized method that has led to uniform application research, education, and clinical practice. EFT is a brief intervention that combines exposure, cognitive therapy, and somatic stimulation of acupressure points on the face and body. It has been reported in the literature that EFT, a "needle-free and emotional" form of acupuncture, reduces or eliminates dysmenorrhea symptoms and premenstrual complaints.

ELIGIBILITY:
Inclusion Criteria:

* • Being a female student at Karabük University Faculty of Health Sciences

  * Being between the ages of 18-25
  * Voluntarily agrees to participate in the study,
  * T.R. to be a citizen,
  * Not having any chronic disease,
  * Those whose symptom complaints are 5 or above according to the VAS scale

Exclusion Criteria:

* • Leaving the study at any time,

  * Having any diagnosed psychiatric disorder.
  * Not having secondary dysmenorrhea pathology

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women
Enrollment: 65 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Examining the Effect of Emotional Freedom Technique on Quality of Life and Symptoms in Dysmenorrhea | Preliminary tests will be carried out and then the 1st EFT session will be held. After 30 days, the first final tests will be performed and then the second EFT session will be held. After 30 days, only the 2nd final tests will be performed.
  Emotional Freedom Technique

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Karabuk University, Karabük, Karabük Province
  - Karabük University, Karabük

IPD SHARING:
Plan to Share IPD: Undecided